CLINICAL TRIAL: NCT04147325
Title: Virologic Response at 48 th Week, in Patients Newly Diagnosed With HIV-1, After the Implementation of a Test and Treat Model of Care, in a Single Portuguese Center.
Brief Title: A Study to Evaluate Virologic Response in Participants Newly Diagnosed With HIV-1
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Farmaceutica Ltda. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108626; TMC114HTX4016 (Other: Janssen-Cilag Farmaceutica Ltda.)
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: HIV
MeSH Terms: interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Participants newly diagnosed with Human Immunodeficiency Virus (HIV)-1, will receive Antiretroviral Therapy (ART) in accordance with clinical practice and will be included in a Test and Treat model of care at the outpatient clinic of the center.
  Interventions: Drug: Antiretroviral Therapy
- Historical Cohort: Naive HIV-1 infected participants who had their first care visit at the outpatient clinic of the center through 2017 will be included in this cohort.
  Interventions: Drug: Antiretroviral Therapy

INTERVENTIONS:
Drug: Antiretroviral Therapy — ART will be administered chosen by the investigator according to country/ local standards/ guidelines/ available ARV for current treatment guidelines for rapid initiation.

SUMMARY:
The purpose of this study is to determine the proportion of newly diagnosed participants with Human Immunodeficiency Virus (HIV)-1 (naive participants) with virologic response at Week 48-defined as HIV-1 Ribonucleic acid (RNA) less than (<) 50 copies/milliliter (mL) (Food And Drug Administration snapshot) - after the implementation of the Test & Treat model of care and in a historical cohort.

ELIGIBILITY:
Inclusion Criteria:

* Prospective cohort: Newly diagnosed with Human Immunodeficiency Virus (HIV)-1 evidenced by any of the following: or HIV Rapid Antibody positive; HIV Immunoassay positive; positive HIV (p24) antigen; or detectable HIV-1 Ribonucleic acid (RNA) Viral Load and non-reactive antibody/antigen assays. HIV-1 RNA Viral Load must be confirmed within one week of initial HIV-1 RNA Viral Load test
* Prospective cohort: Antiretroviral (ARV) treatment-naïve who will initiate treatment. Retrospective cohort: Dates of HIV-1 diagnosis and ARV treatment initiation available in clinical records
* Prospective and Retrospective cohorts: Must sign [and/or their legally-acceptable representative where applicable must sign,] a participation agreement/ Informed Consent Form (ICF) allowing data collection and source data verification in accordance with local requirements

Exclusion Criteria:

* Known Acquired Immune Deficiency Syndrome (AIDS)-defining condition
* Known history of clinically relevant hepatic disease or hepatitis that in the investigator's judgement is not compatible with Antiretroviral Therapy (ART)
* Known history of chronic renal insufficiency, defined as having an eGFR less than (<) 50 milliliter/minute (ml/min) according to the Cockcroft-Gault formula
* Known active severe infections (other than HIV-1 infection) requiring parenteral antibiotic or antifungal therapy within 30 days prior to screening
* Known history of cirrhosis as diagnosed based on local practices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants newly diagnosed with Human Immunodeficiency Virus (HIV)-1, who will be included in a Test and Treat model of care (Prospective Cohort) and naive HIV-infected participants who had their first care visit at the outpatient clinic of the center through 2017 (Retrospective Cohort) will be observed. Only data available as per clinical practice will be collected within this study.
Sampling Method: Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Percentage of Newly Diagnosed Participants with Human Immunodeficiency Virus (HIV)-1 Ribonucleic acid (RNA) < 50 Copies per Milliliter (c/mL) at Week 48 (Virologic Response) | Week 48
  The percentage of newly diagnosed participants is defined as the percentage of newly HIV-1 infected participants that are considered virologic responders (that is have HIV-1 RNA viral load less than [<] 50 c/mL) at Week 48 as per the Food And Drug Administration (FDA) snapshot algorithm.

SECONDARY OUTCOMES:
Time to Antiretroviral Therapy (ART) Initiation since HIV-1 Diagnosis | Up to 48 weeks
  Time to ART initiation is defined as time from HIV diagnosis (date of the first HIV positive test) to the start of ART.
Time to Virologic Suppression | Up to 48 weeks
  Time to virologic suppression is defined as time from start of ART to the HIV RNA < 50 copies/mL measured as per FDA snapshot algorithm.
Time to Virologic Response | Up to 48 weeks
  Time to virologic response is defined as HIV-1 RNA viral load (VL) < 200 copies/mL measured as per FDA snapshot algorithm.
Change from Baseline in HIV-1 RNA from Start of ART | Baseline up to week 48
  Change from baseline in HIV-1 RNA will be assessed through time (up to Week 48) from the date of start of ART.
Change from Baseline in Cluster Differentiation 4 (CD4) Cell Count | Baseline up to Week 48
  Change from baseline in CD4 cell count for immunologic changes after ART initiation will be determined.
Change from Baseline in Viral Load | Baseline up to Week 48
  Change from baseline in viral load for virologic changes after ART initiation will be determined.
Percentage of Participants not Lost-to-Follow up | 12 months
  The percentage of participants who maintained regular visits to the HIV center during a 12-month period after HIV diagnose period will be reported.
Time from HIV Diagnosis to First Care Visit | Baseline (Day 1)
  Time from HIV diagnosis to first care visit will be performed by evaluating time between diagnosis of HIV and date of the first care visit.
Time from First Care Visit to ART Initiation | Baseline (Day 1)
  Time from first care visit to ART initiation in all newly diagnosed patients with HIV will be reported.
Percentage of Participants Developing PR, RT, and INI Resistance-Associated Mutation (RAMs) During Follow-up | Through 4, 6, 12, 24 and 48 weeks
  Percentage of participants developing protease (PR), reverse transcriptase (RT), and integrase (INI) RAMs during follow-up will be reported.
Percentage of Participants who Loss-to-Follow According to Burkitt lymphoma (BL) CD4 cell Count | Up to 24 Months (end of study)
  Percentage of participants who lost-to-follow up according to BL CD4 cell count, in all newly diagnosed participants with HIV will be reported.
Change from Baseline in ARV Regimen due to Resistance | Baseline up to Week 48
  Changes from baseline in ARV regimen due to resistance, will be evaluated in all newly diagnosed participants with HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Farmaceutica Ltda. Clinical Trial, Study Director — Janssen-Cilag Farmaceutica Ltda.
Locations (1):
- Chlo - Hosp. Egas Moniz, Lisbon, Portugal

IPD SHARING:
Plan to Share IPD: No